CLINICAL TRIAL: NCT02493647
Title: Reducing Urban Women's HIV Risk: Soap Opera Videos on Mobile Devices
Brief Title: Love, Sex & Choices: A Web Series on Mobile Devices to Reduce Black Women's HIV Risk
Acronym: LSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northeastern University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Rachel Jones, RN, PhD, Associate Professor, Northeastern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LSCR012015; 1R01NR014632 (NIH)
Record Dates: First submitted 2015-06-24; First posted 2015-07-09 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: HIV; Sexual Behavior; Women's Role; Risk Behavior; Chlamydia
MeSH Terms: conditions — Sexual Behavior; Risk-Taking; Chlamydia Infections | interventions — Sex

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Love, Sex, & Choices (Experimental): Love, Sex, and Choices (LSC) is an engaging 12-episode video series to reduce HIV risk in young, adult predominately Black women. A peer video guide was added to the end of LSC episodes to provoke viewers to question their own sex scripts and consider their own need for change. Investigators propose to conduct a two-arm clinical trial of guide enhanced LSC impact on reducing unprotected sex with high risk partners and increasing HIV testing in Black women in high HIV prevalence neighborhoods.
  Interventions: Behavioral: Love, Sex, & Choices
- Attention-Time Control (No Intervention): The Control is a 12-episode popular web miniseries with a storyline that promotes respectful relationships. time and frequency are matched to the active intervention.

INTERVENTIONS:
Behavioral: Love, Sex, & Choices — Investigators propose to conduct a two-arm clinical trial of guide enhanced LSC impact on reducing unprotected sex with high risk partners and increasing HIV testing in Black women in high HIV prevalence neighborhoods. Undiagnosed HIV is a significant factor fueling the epidemic. Recruitment into the study will be via Facebook or traditional on the ground.
  Other Names: guide enhanced Love, Sex, & Choices
  Arms: Love, Sex, & Choices

SUMMARY:
This study tests a 12-episode Internet-based, guide enhanced Love, Sex, & Choices (LSC) HIV prevention soap opera video series for smartphones or computers, in a randomized clinical trial among predominately at-risk African American urban women.

The following hypotheses are to be tested: 1) The LSC treatment arm will show lower unprotected sex risk, meaning lower frequency of unprotected sex (vaginal + anal) with high risk partners at 6 months post intervention compared to an attention control arm 2) The LSC treatment arm will show higher participation in HIV testing at 6 months post intervention compared to the control.

If effective, this video intervention could be rapidly implemented and brought to scale at low cost via the Internet, widely reaching young urban women with the goal of reducing HIV risk behavior and increasing HIV testing.

DETAILED DESCRIPTION:
Love, Sex, and Choices (LSC) is an engaging 12-episode video series to reduce HIV risk in young, adult predominately Black women. A peer video guide was added to the end of LSC episodes to provoke viewers to question their own sex scripts and consider their own need for change. The investigators propose to conduct a two-arm clinical trial of the guide enhanced LSC impact on reducing unprotected sex with high risk partners and increasing HIV testing in Black women in high HIV prevalence neighborhoods. Undiagnosed HIV is a significant factor fueling the epidemic. The Control is a 12-episode popular web miniseries with a storyline that promotes respectful relationships. A previous online pilot study was conducted to evaluate the guide enhanced LSC acceptability, the feasibility of Facebook® advertising, and streaming the guide enhanced LSC to smartphones. This pilot study indicated 43.6% went for HIV testing within 30 days post viewing. The guide enhanced LSC was associated with sex risk reduction. Recruitment and retention of Black women in online HIV prevention research remain understudied.

AIM 1 is to conduct a RCT to evaluate the effect of the guide enhanced LSC on HIV sex risk behavior compared to a true attention control.

AIM 2 is to evaluate effect of the guide enhanced LSC on HIV testing. AIM 3 is to compare the reach, meaning enrollment, engagement, retention, risk behaviors, and demographics of high risk, young urban Black women recruited online to those obtained by conventional recruitment: with and without research team assistance, to determine whether online recruitment reaches subgroups not reached in conventional recruitment. Data from Facebook© ads, QR codes, site specific URL on flyers, tracking video viewing, retention data, and risk behaviors will help evaluate efforts to reach and retain high risk women.

AIM 4 is to specify a model of the effect of the guide enhanced LSC series on high risk sex scripts and sex risk. Storytelling can promote behavior change but the study of the mechanism of effect is still young, and entertainment-education concepts of effective film are not yet well integrated into HIV prevention science. Identification with film characters and transportation, characterized by emotional and cognitive empathy and merging, are known to mediate cognitive shifts.

The following hypotheses are to be tested in a RCT in predominately young urban Black women [1) The guide enhanced LSC treatment arm will show lower unprotected sex risk, meaning lower frequency of unprotected sex (vaginal + anal) with high risk partners at 6 months post intervention compared to an attention control arm (2) The guide enhanced LSC treatment arm will show higher participation in HIV testing at 6 months post intervention compared to the control. Investigators will learn by secondary analyses, whether (3) there are differences in reach by Facebook© compared to conventional recruitment, and 4) Retention of at risk women recruited online will be similar to those recruited in the field and 5) whether identification and transportation will lower high risk sex scripts as a mediator of lower USR and greater HIV testing.

ELIGIBILITY:
Inclusion Criteria:

* sexual relationship with a man in previous 3 months
* speak and read English

Exclusion Criteria:

* younger than 18 years old
* older than 29 years old
* currently pregnant
* women who have already participated in the study

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 814 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Frequency of unprotected vaginal or anal sex with perceived high risk male partner | 6 months
  test hypothesis that the LSC treatment arm will show lower unprotected sex risk, meaning lower frequency of unprotected sex (vaginal + anal) with high risk partners at 6 months post intervention compared to an attention control arm
Incidence of HIV testing | 6 months
  Test hypothesis that the LSC treatment arm will show higher participation in HIV testing at 6 months post intervention compared to the control

SECONDARY OUTCOMES:
composite demographic measure | 6 months
  test whether there are differences in demographics between recruitment online on Facebook© compared to conventional recruitment
Attrition | 6 months
  test whether there are differences in those who do not complete the study between recruitment online on Facebook© compared to conventional recruitment
Identification with Character Scale | 1 month
  test whether identification and transportation will lower high risk sex scripts as a mediator of reducing sex risk and increased HIV testing.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Jones, PhD, Principal Investigator — Northeastern University
Locations (1):
- Northeastern University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No